CLINICAL TRIAL: NCT05202093
Title: Efficacy of Two Sonic Toothbrushes in Reducing Extrinsic Tooth Stain: An 8-week Randomized Clinical Trial
Brief Title: Efficacy of Two Sonic Toothbrushes in Reducing Extrinsic Tooth Stain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Liu Hongchun, Principal Investigator, Hospital of Stomatology, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Whitening sonic toothbrush
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Results first posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Tooth Bleaching
Keywords: Controlled Clinical Trial; Electric Toothbrush

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- the Oclean Digital Visual toothbrush (2.16 N·cm torque) (Experimental): Use the Oclean Digital Visual toothbrush (2.16 N·cm torque) to brush teeth twice daily for 8 weeks
  Interventions: Device: the Oclean Digital Visual toothbrush (2.16 N·cm torque)
- the Oclean Sonic Electric toothbrush (1.96 N·cm torque) (Experimental): Use the Oclean Sonic Electric toothbrush (1.96 N·cm torque) to brush teeth twice daily for 8 week
  Interventions: Device: the Oclean Sonic Electric toothbrush (1.96 N·cm torque)
- Manual toothbrush (Active Comparator): Use Oral-B manual toothbrush to brush teeth twice daily for 8 weeks
  Interventions: Device: Oral B manual toothbrush

INTERVENTIONS:
Device: the Oclean Digital Visual toothbrush (2.16 N·cm torque) — Use the Oclean Digital Visual toothbrush (2.16 N·cm torque) to brush teeth twice a day for 8 weeks
  Arms: the Oclean Digital Visual toothbrush (2.16 N·cm torque)
Device: Oral B manual toothbrush — Use Oral B manual toothbrush to brush teeth twice a day for 8 weeks
  Arms: Manual toothbrush
Device: the Oclean Sonic Electric toothbrush (1.96 N·cm torque) — Use the Oclean Sonic Electric toothbrush (1.96 N·cm torque) to brush teeth twice a day for 8 weeks
  Arms: the Oclean Sonic Electric toothbrush (1.96 N·cm torque)

SUMMARY:
The objective of the present study was to compare the effects of reduction of extrinsic stains between 2 commercially available Oclean sonic toothbrushes in comparison with an Oral-B manual toothbrush.

DETAILED DESCRIPTION:
Extrinsic tooth stain, especially on anterior teeth, is a common aesthetic issue that affect smile and self-confidence. Epidemiological studies show that dissatisfaction with tooth color impacts approximately 20% to 60% of various population groups. In a Chinese urban sample, 52.6% reported dissatisfaction with tooth color. Patients often express a desire to achieve whiter teeth, as it improves smile aesthetics, attractiveness and quality of life. It also promotes overall oral health and well-being.

Mechanical tooth cleaning through brushing remains the most effective approach for daily oral hygiene, effectively removing plaque and stain to maintain oral health, irrespective of the use of dentifrice. The effectiveness of manual toothbrush is predominantly influenced by users' brushing habits and their compliance with professional recommendations.

The electric toothbrush was first introduced in Switzerland in 1954. It was designed to simulate and enhance manual brushing motions, thereby potentially offering an improved cleaning experience. Modern electric toothbrushes feature integrated timers, pressure sensors, multiple brushing modes, and Bluetooth-enabled apps to enhance brushing duration and quality. The Oclean Digital Visual toothbrush and Oclean Sonic Electric toothbrush, developed by a Shenzhen-based Chinese company, exemplify these innovations. Both sonic toothbrushes feature silent motor technology to reduce noise, avoid resonant frequencies to lessen facial discomfort, and provide real-time pressure feedback to prevent excessive brushing force. Together, these enhancements ensure a quieter, smoother, and more comfortable brushing experience. While both models share core manufacturing parameters, the Oclean Digital Visual toothbrush provides a higher driving torque (2.16 N.cm) than the Oclean Sonic Electric toothbrush (1.96 N.cm).

ELIGIBILITY:
The inclusion criteria were: 1) aged 18-70 years; 2) good general health; 3) ability to attend all scheduled visits over the 8-week study period; 4) possession of more than 20 natural permanent teeth, excluding third molars, which are free of crowns or extensive restorative materials; 5) at least 12 anterior teeth suitable for scoring (i.e., free of crowns, veneers, large restorations, trauma, or non-vital pulp); 6) a whole-mouth mean Lobene stain composite score greater than 1.

Exclusion criteria included: 1) severe oral or systemic diseases; 2) advanced periodontal diseases; 3) pregnancy or lactation; 4) dental fluorosis or tetracycline staining; 5) orthodontic appliances or partial removable dentures; 6) participation in other clinical trials; 7) professional prophylaxis within 3 months or tooth whitening within 6 months; and 8) known allergy to study products.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-03-05 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hongchun Liu, Principal Investigator — Guanghua School of Stomatology, Sun Yat-sen University
Locations (1):
- Hongchun Liu, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- the Oclean Digital Visual Toothbrush (2.16 N·cm Torque): Use the Oclean Digital Visual toothbrush (2.16 N·cm torque) to brush teeth twice daily for 8 weeks
  Oclean electric toothbrush A: Use the Oclean Digital Visual toothbrush (2.16 N·cm torque)to brush teeth twice a day for 8 weeks
- the Oclean Sonic Electric Toothbrush (1.96 N·cm Torque): Use the Oclean Sonic Electric toothbrush (1.96 N·cm torque) to brush teeth twice daily for 8 week
  Oclean electric toothbrush B: Usethe Oclean Sonic Electric toothbrush (1.96 N·cm torque) to brush teeth twice a day for 8 weeks
- Manual Toothbrush: Use Oral-B manual toothbrush to brush teeth twice daily for 8 weeks
  Oral-B manual toothbrush: Use Oral B manual toothbrush to brush teeth twice a day for 8 weeks
Period: Overall Study
Arm/Group | the Oclean Digital Visual Toothbrush (2.16 N·cm Torque) | the Oclean Sonic Electric Toothbrush (1.96 N·cm Torque) | Manual Toothbrush
Started | 43 | 43 | 43
Completed | 43 | 42 | 41
Not Completed | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- the Oclean Digital Visual Toothbrush (2.16 N·cm Torque): Use the Oclean Digital Visual toothbrush (2.16 N·cm torque) to brush teeth twice daily for 8 weeks
  Oclean the Oclean Digital Visual toothbrush (2.16 N·cm torque) : Use the Oclean Digital Visual toothbrush (2.16 N·cm torque) to brush teeth twice a day for 8 weeks
- the Oclean Sonic Electric Toothbrush (1.96 N·cm Torque): Use the Oclean Sonic Electric toothbrush (1.96 N·cm torque) to brush teeth twice daily for 8 week
  Oclean the Oclean Sonic Electric toothbrush (1.96 N·cm torque): Use the Oclean Sonic Electric toothbrush (1.96 N·cm torque) to brush teeth twice a day for 8 weeks
- Total: Total of all reporting groups
Arm/Group | the Oclean Digital Visual Toothbrush (2.16 N·cm Torque) | the Oclean Sonic Electric Toothbrush (1.96 N·cm Torque) | Manual Toothbrush | Total
Number analyzed (Participants) | 43 | 42 | 41 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.02 (8.87) | 43.98 (9.98) | 44.15 (8.28) | 43.71 (9.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 24 | 76
  Male | 17 | 16 | 17 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Han | 43 | 42 | 41 | 126
Lobene Stain Index of Stain Intensity Scores [Mean (Standard Deviation); unit: score on a scale] — Each tooth surface was divided into two regions: body and gingival. For each region, tooth stain intensity was rated on a 0-3 ordinal scale (minimum = 0, maximum = 3),using the Lobene Stain Index: 0 = No stain; 1 = Light stain (yellow to light brown or gray); 2 = Moderate stain (medium brown); 3 = Heavy stain (dark brown to black).
  The mean Lobene stain intensity score was calculated by summing the scores from all assessed regions of the tooth surfaces and dividing by the total number of regions.
  Higher scores indicate a worse outcome (i.e., more severe extrinsic tooth stain).
  score on a scale | 1.28 (0.48) | 1.28 (0.57) | 1.31 (0.52) | 1.29 (0.52)
Lobene Stain Index of Stain Area Scores [Mean (Standard Deviation); unit: score on a scale] — Each tooth surface was divided into two regions: body and gingival. For each region, tooth stain area was rated on a 0-3 ordinal scale (minimum = 0, maximum = 3), using the Lobene Stain Index: 0= no stain detected; 1= stain covering up to 1/3 of the region; 2= stain covering >1/3 to 2/3 of the region; 3=stain covering >2/3 of the region.
  The mean Lobene stain area score was calculated by summing the scores from all assessed regions of the tooth surfaces and dividing by the total number of regions.
  Higher scores indicate a worse outcome (i.e., more severe extrinsic tooth stain).
  score on a scale | 1.1 (0.35) | 1.13 (0.43) | 1.14 (0.39) | 1.12 (0.39)
Lobene Stain Index of Stain Composite Scores [Mean (Standard Deviation); unit: score on a scale] — Each tooth surface was divided into two regions: body and gingival. For each region, a composite score is calculated by averaging the product of the intensity and extent scores.
  Each subscale (body and gingival) has a range of 0-9 (minimum = 0, maximum = 9).
  The mean Lobene stain composite score was determined by summing the scores from all assessed regions of the tooth surfaces and dividing by the total number of regions evaluated.
  Higher scores indicate a worse outcome (i.e., more severe extrinsic tooth stain).
  score on a scale | 2.4 (1.03) | 2.35 (1.24) | 2.37 (1.16) | 2.37 (1.13)

OUTCOME MEASURES:

1. Primary Outcome: Lobene Stain Index of Stain Intensity Scores 4 Weeks After Toothbrush Use
Description: Tooth stain of the anterior teeth was measured using the Lobene Stain Index. The index assesses the area and intensity of extrinsic tooth stain on the facial and lingual surfaces of the lower anterior teeth and the facial surfaces of the upper anterior teeth. Each evaluated tooth surface was divided into two anatomical regions: body and gingival. For each region, stain intensity was rated on a 0-3 ordinal scale with the following criteria: 0 = No stain; 1 = Light stain (yellow to light brown or gray); 2 = Moderate stain (medium brown); 3 = Heavy stain (dark brown to black).
  Each region(body and gingival) has a score range of 0-3 (minimum = 0, maximum = 3).
  The mean Lobene stain intensity score was determined by summing the scores from all assessed regions of the tooth surfaces and dividing by the total number of regions evaluated.
  Higher scores (both subscale and mean score) indicate a worse outcome (i.e., more severe extrinsic tooth stain).
Time Frame: 4 weeks after toothbrush use
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- the Oclean Digital Visual Toothbrush (2.16 N·cm Torque): Use the Oclean Digital Visual toothbrush (2.16 N·cm torque) to brush teeth twice daily for 8 weeks
  the Oclean Digital Visual toothbrush (2.16 N·cm torque) : Use Oclean electric toothbrush A to brush teeth twice a day for 8 weeks
- the Oclean Sonic Electric Toothbrush (1.96 N·cm Torque): Use the Oclean Sonic Electric toothbrush (1.96 N·cm torque) to brush teeth twice daily for 8 week
  the Oclean Sonic Electric toothbrush (1.96 N·cm torque): Use Oclean electric toothbrush B to brush teeth twice a day for 8 weeks
Arm/Group | the Oclean Digital Visual Toothbrush (2.16 N·cm Torque) | the Oclean Sonic Electric Toothbrush (1.96 N·cm Torque) | Manual Toothbrush
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 0.89 (0.48) | 0.88 (0.46) | 1.13 (0.55)

2. Primary Outcome: Lobene Stain Index of Stain Area Scores 4 Weeks After Toothbrush Use
Description: Tooth stain of the anterior teeth was measured using the Lobene Stain Index. The index assesses the area and intensity of extrinsic tooth stain on the facial and lingual surfaces of the lower anterior teeth and the facial surfaces of the upper anterior teeth. Each evaluated tooth surface was divided into two anatomical regions: body and gingival. For each region, the stain area score were assessed using 0-3 scale. 0= no stain detected; 1= stain covering up to 1/3 of the region; 2= stain covering >1/3 to 2/3 of the region; 3=stain covering >2/3 of the region.
  Each region (body and gingival) has a score range of 0-3 (minimum = 0, maximum = 3).
  The mean Lobene stain area score was determined by summing the scores from all assessed regions of the tooth surfaces and dividing by the total number of regions evaluated.
  Higher scores (both subscale and mean score) indicate a worse outcome (i.e., more severe extrinsic tooth stain).
Time Frame: 4 weeks after toothbrush use
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- the Oclean Sonic Electric Toothbrush (1.96 N·cm Torque): Use the Oclean Sonic Electric toothbrush (1.96 N·cm torque)to brush teeth twice daily for 8 week
  the Oclean Sonic Electric toothbrush (1.96 N·cm torque): Use the Oclean Sonic Electric toothbrush (1.96 N·cm torque) to brush teeth twice a day for 8 weeks
Arm/Group | the Oclean Digital Visual Toothbrush (2.16 N·cm Torque) | the Oclean Sonic Electric Toothbrush (1.96 N·cm Torque) | Manual Toothbrush
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 0.81 (0.37) | 0.81 (0.43) | 1.02 (0.43)

3. Primary Outcome: Lobene Stain Index of Stain Composite Scores 4 Weeks After Toothbrush Use
Description: Tooth stain of the anterior teeth was measured using the Lobene Stain Index. The index assesses the area and intensity of extrinsic tooth stain on the facial and lingual surfaces of the lower anterior teeth and the facial surfaces of the upper anterior teeth. Each evaluated tooth surface was divided into two anatomical regions: body and gingival. For each region, a composite score is calculated by averaging the product of the intensity and extent scores.
  Each region (body and gingival) has a score range of 0-9 (minimum = 0, maximum = 9).
  The mean Lobene stain composite score was determined by summing the scores from all assessed regions of the tooth surfaces and dividing by the total number of regions evaluated.
  Higher scores (both subscale and mean score) indicate a worse outcome (i.e., more severe extrinsic tooth stain).
Time Frame: 4 weeks after toothbrush use
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- the Oclean Sonic Electric Toothbrush (1.96 N·cm Torque): Use the Oclean Sonic Electric toothbrush (1.96 N·cm torque) to brush teeth twice daily for 8 week
  the Oclean Sonic Electric toothbrush (1.96 N·cm torque): Use the Oclean Sonic Electric toothbrush (1.96 N·cm torque)B to brush teeth twice a day for 8 weeks
Arm/Group | the Oclean Digital Visual Toothbrush (2.16 N·cm Torque) | the Oclean Sonic Electric Toothbrush (1.96 N·cm Torque) | Manual Toothbrush
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 1.54 (0.94) | 1.5 (0.96) | 2.05 (1.21)

4. Primary Outcome: Lobene Stain Index of Stain Intensity Scores 8 Weeks After Toothbrush Use
Description: as for outcome 1
Time Frame: 8 weeks after toothbrush use
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- the Oclean Digital Visual Toothbrush (2.16 N·cm Torque): Use the Oclean Digital Visual toothbrush (2.16 N·cm torque)to brush teeth twice daily for 8 weeks
  the Oclean Digital Visual toothbrush (2.16 N·cm torque): Usethe Oclean Digital Visual toothbrush (2.16 N·cm torque) to brush teeth twice a day for 8 weeks
Arm/Group | the Oclean Digital Visual Toothbrush (2.16 N·cm Torque) | the Oclean Sonic Electric Toothbrush (1.96 N·cm Torque) | Manual Toothbrush
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 0.78 (0.41) | 0.71 (0.4) | 1.01 (0.52)

5. Primary Outcome: Lobene Stain Index of Stain Area Scores 8 Weeks After Toothbrush Use
Description: as for outcome 2
Time Frame: 8 weeks after toothbrush use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | the Oclean Digital Visual Toothbrush (2.16 N·cm Torque) | the Oclean Sonic Electric Toothbrush (1.96 N·cm Torque) | Manual Toothbrush
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 0.75 (0.33) | 0.74 (0.42) | 0.94 (0.45)

6. Primary Outcome: Lobene Stain Index of Stain Composite Scores 8 Weeks After Toothbrush Use
Description: as for outcome 3
Time Frame: 8 weeks after toothbrush use
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | the Oclean Digital Visual Toothbrush (2.16 N·cm Torque) | the Oclean Sonic Electric Toothbrush (1.96 N·cm Torque) | Manual Toothbrush
Number analyzed (Participants) | 43 | 42 | 41
score on a scale | 1.37 (0.87) | 1.27 (0.84) | 1.88 (1.21)

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- the Oclean Digital Visual Toothbrush (2.16 N·cm Torque): Use the Oclean Digital Visual toothbrush (2.16 N·cm torque) to brush teeth twice daily for 8 weeks
  Oclean electric toothbrush A: Use the Oclean Digital Visual toothbrush (2.16 N·cm torque) to brush teeth twice a day for 8 weeks
Arm/Group | the Oclean Digital Visual Toothbrush (2.16 N·cm Torque) | the Oclean Sonic Electric Toothbrush (1.96 N·cm Torque) | Manual Toothbrush
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/42 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/41
Other Adverse Events (participants affected / at risk) | 0/43 | 0/42 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT05202093/Prot_SAP_000.pdf